CLINICAL TRIAL: NCT07255807
Title: sIgnatuRe: Defining the Human Insulin Resistance Molecular Network
Brief Title: Defining the Human Insulin Resistance Molecular Network; SIGNATURE
Acronym: SIGNATURE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: University of Sydney (Other); Queen Mary University of London (Other); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Jorgen FP Wojtaszewski, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SIGNATURE; NNF24OC0085866 (Other Grant/Funding Number: Novo Nordisk Foundation)
Record Dates: First submitted 2025-08-06; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Metabolic Health; Insulin Sensitivity/Resistance
Keywords: Insulin Resistance; Metabolic Health; Glucose Metabolism; Lifestyle Interventions; Physical Inactivity; High-Fat Diet; Molecular Mechanisms; Insulin Sensitivity; Metabolic Phenotyping; Human Intervention Study
MeSH Terms: conditions — Insulin Resistance; Sedentary Behavior | interventions — Parenteral Nutrition

STUDY DESIGN:
Intervention Model Description: This study uses a parallel design involving 80 healthy participants who all undergo comprehensive baseline assessments, including physiological and metabolic phenotyping, habitual physical activity, and dietary intake evaluations. Following baseline characterization, 40 participants are assigned to one of two independent intervention arms: 14 days of reduced physical activity or 3 days of a hypercaloric high-fat diet. Each intervention group is studied in parallel, with outcomes compared to assess the specific effects on insulin sensitivity and molecular mechanisms. The parallel design was chosen due to the invasive and time-intensive nature of the interventions and testing procedures, making a crossover design impractical and burdensome for participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline Characterization (No Intervention): All participants (N=80) undergo extensive baseline characterization over three study visits. This includes assessments of insulin sensitivity, glucose tolerance, metabolic and physiological phenotyping, habitual physical activity, and dietary intake. No intervention is applied during this phase; the purpose is to establish baseline measures and characterize individual variation in insulin resistance and metabolic profiles.
  Participants complete detailed clinical, physiological, and behavioral assessments without any experimental manipulation. This includes:
  * Measurement of insulin action and glucose tolerance
  * Dietary and physical activity profiling
  * Collection of biospecimens for molecular analyses
- Lifestyle Interventions (Experimental): A subset of 40 participants are randomized into one of two experimental interventions following baseline assessment:
  * 14 days of reduced physical activity (<1,500 steps/day), or
  * 3 days of a hypercaloric high-fat diet
  The aim is to evaluate how short-term lifestyle stressors affect insulin sensitivity and related molecular markers. Assessments from visits 4 and 5 are compared to baseline to determine within-subject changes.
  Intervention Names:
  1. Reduced Physical Activity
     - Participants limit daily steps to <1,500 for 14 days
  2. High-Fat Diet
     * Participants consume a hypercaloric, high-fat diet for 3 days
  Description of Intervention:
  Participants undergo one of the two lifestyle interventions with strict monitoring and support. Selected baseline tests are repeated post-intervention to evaluate metabolic and molecular responses.
  Interventions: Behavioral: Physical Inactivity; Behavioral: Hypercaloric High-Fat Diet

INTERVENTIONS:
Behavioral: Physical Inactivity — Participants assigned to the physical inactivity intervention will reduce their daily physical activity to fewer than 1,500 steps per day for 14 consecutive days. This strict limitation significantly decreases overall movement and muscle activity, mimicking a sedentary lifestyle. The aim is to assess the short-term effects of reduced physical activity on insulin sensitivity and related metabolic processes. Compliance will be monitored using activity trackers and daily logs. Baseline metabolic and physiological assessments will be repeated after the intervention to evaluate changes.
  Other Names: Reduced Activity
  Arms: Lifestyle Interventions
Behavioral: Hypercaloric High-Fat Diet — Participants assigned to the high-fat diet intervention will consume a hypercaloric diet rich in fat for 3 consecutive days. The diet is designed to significantly increase caloric intake and fat consumption beyond habitual levels to induce short-term metabolic stress. This intervention aims to assess how a brief period of high-fat overfeeding affects insulin sensitivity and related molecular pathways. Participants' dietary intake will be carefully controlled and monitored to ensure adherence. Baseline metabolic and physiological assessments will be repeated after the intervention to evaluate changes.
  Other Names: Overeating
  Arms: Lifestyle Interventions

SUMMARY:
The goal of this intervention study is to learn more about what causes insulin resistance in otherwise healthy adults, and how short-term changes in physical activity or diet may influence it. The study includes healthy male and female participants aged 25 to 55 years, who meet specific health criteria.

The main questions it aims to answer are:

Does the cause of insulin resistance vary between individuals due to their genes and lifestyle?

Can the investigators identify different types (sub-phenotypes) of insulin resistance at the molecular level?

Researchers will compare groups who either reduce their physical activity for 14 days or consume a high-fat diet for 3 days, to see how these changes affect insulin sensitivity and related biological markers.

Participants will:

* Complete a health screening and be assessed for eligibility
* Undergo baseline testing to measure insulin sensitivity, physical activity, diet, and metabolic health
* Be randomly assigned to one of two short-term interventions (14 days of reduced physical activity, or 3 days of a high-fat, high-calorie diet)
* Repeat selected tests after the intervention to assess changes

This study will help researchers better understand how lifestyle and biology interact in the development of insulin resistance, even in people who are otherwise healthy.

DETAILED DESCRIPTION:
This intervention study aims to uncover the molecular mechanisms that underlie insulin resistance in otherwise healthy adults and to explore how short-term lifestyle changes may influence these mechanisms. Insulin resistance is a key feature in the development of type 2 diabetes and other metabolic diseases, but it does not arise uniformly across individuals. The overarching hypothesis is that insulin resistance has multiple underlying causes that differ between individuals, depending on genetic variation and modifiable lifestyle factors such as physical activity and diet.

A total of 80 healthy participants-40 males and 40 females aged between 25 and 55 years-will be recruited. All participants must have a body mass index (BMI) between 18 and 30 and meet strict inclusion and exclusion criteria to minimize confounding variables. Participants will be free of chronic disease, non-smokers, have limited alcohol intake, and not engage in high levels of physical activity. This controlled approach ensures a more accurate assessment of the variables under investigation.

At baseline, all participants will undergo comprehensive phenotyping, including assessments of habitual physical activity, dietary intake, glucose tolerance, and whole-body insulin sensitivity. This will allow the researchers to categorize sub-phenotypes of insulin resistance at both the physiological and molecular level.

Following baseline testing, 40 of the 80 participants will undergo one of two short-term interventions designed to stress metabolic pathways associated with insulin sensitivity:

* Reduced physical activity: Participants will significantly decrease their daily physical activity for 14 days.
* High-fat diet: Participants will consume a hypercaloric high-fat diet for 3 consecutive days.

The aim of these interventions is to test how short-term negative lifestyle changes impact insulin action and related molecular markers, and whether these responses vary between individuals with different phenotypic and genetic profiles.

After the intervention period, selected metabolic tests will be repeated to assess changes in insulin sensitivity and molecular signaling. The primary outcome measure is whole-body insulin action, assessed using gold-standard physiological methods. Exploratory outcomes include identifying cellular and molecular mechanisms contributing to insulin resistance, and understanding the interaction between gene expression and lifestyle responses.

By combining deep phenotyping with short-term interventions, this study will generate new insights into the biological diversity of insulin resistance. Ultimately, this may contribute to the development of more individualized strategies for the prevention and treatment of metabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25-55 years
* Body Mass Index (BMI): 18-30 kg/m²
* Healthy (no diagnosed chronic diseases)
* Able and willing to comply with study procedures

Exclusion Criteria:

* Smoking or nicotine use, current or within the past 5 years
* Alcohol intake exceeding 10 units per week
* Hemoglobin A1c (HbA1c) > 48 mmol/mol (indicative of diabetes or prediabetes)
* Chronic diseases (e.g., cardiovascular disease, diabetes, etc.)
* Chronic medication use, including hormonal treatments
* High physical activity levels (more than 3 hours per week of moderate to vigorous exercise)
* Pregnancy or within 3 months postpartum
* Breastfeeding or within 3 months of cessation
* Abnormal routine blood markers (as defined in lab screening)
* Blood donation within the past 2 months

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2038-06-30 (Estimated)

PRIMARY OUTCOMES:
Whole-body insulin action | Baseline characterization & immediately following intervention (either 14 days of physical inactivity or 3 days of hypercaloric high-fat diet)
  Glucose disposal rates during hyperinsulinemic euglycemic conditions as a marker of whole-body insulin action

SECONDARY OUTCOMES:
Identification of proteins and posttranslational modification of proteins in blood as well as skeletal muscle and adipose tissue biopsies | Baseline & immediately following the intervention (14 days of physical inactivity or 3 days of hypercaloric high-fat diet)
  The obtained skeletal muscle samples will be subjected to mass spectrometry-based proteomic and phosphoproteomic analyses. These measurements show protein abundance and posttranslational modifications that regulates protein function. Ultimately, revealing the signalling network underlying the interventions studied. Unit of measure is log2-transformed arbitrary units.
Whole-Body Glucose Tolerance | Baseline & immediately following the intervention (14 days of physical inactivity or 3 days of hypercaloric high-fat diet)
  Whole-body glucose tolerance will be assessed by an oral glucose tolerance test (OGTT). Blood glucose and insulin concentrations will be measured at multiple time points following oral glucose ingestion to determine glucose and insulin responses. Glucose and insulin areas under the curve (AUC) values will be used to evaluate changes in glucose tolerance.
Beta Cell Function | Baseline & immediately following the intervention (14 days of physical inactivity or 3 days of hypercaloric high-fat diet)
  Beta cell function will be evaluated using an intravenous glucose tolerance test (IVGTT). Following intravenous glucose administration, arterial glucose and insulin concentrations will be measured at multiple time points to assess first-phase insulin secretion and beta cell responsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen F.P. Wojtaszewski, Ph.D., Principal Investigator — University of Copenhagen; Ylva Hellsten, Ph.D., Principal Investigator — University of Copenhagen; Henriette Pilegaard, Ph.D., Principal Investigator — University of Copenhagen
Locations (1):
- August Krogh Building, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the physiological and molecular data collected, and the relatively small and deeply phenotyped cohort, there is a risk of re-identification. Participants have not provided explicit consent for public sharing of their individual data. Furthermore, data protection regulations under the EU General Data Protection Regulation (GDPR) place strict limitations on the sharing of personal data, particularly when it concerns health-related information. For these reasons, individual participant data will not be shared publicly. Data sharing may be considered in the future under controlled access with appropriate ethical approvals and data use agreements.